CLINICAL TRIAL: NCT01619995
Title: Brain Imaging Plus Urodynamics to Investigate the Brain's Control of the Bladder
Acronym: NIRS/fBFB
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Becky Clarkson, Research Instructor in Medicine, University of Pittsburgh
Other Study IDs: PRO10020240; 1R03AG038583-01 (NIH)
Record Dates: First submitted 2012-06-12; First posted 2012-06-15 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Urge Urinary Incontinence
Keywords: urge incontinence
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this project is to evaluate the applicability of non-invasive optical imaging for the measurement of brain function during investigation of the lower urinary tract.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory women over age 60, who are incontinent at least five times weekly for 3 months despite correction of potentially reversible causes.
* urinary incontinence (urge or predominantly urge) by clinical criteria.
* able to accurately complete a voiding diary, to perform a 24-hour pad test under direction.

Exclusion Criteria:

* significant mental impairment [mini mental status exam (MMSE) ≤ 20)
* urethral obstruction
* history of bladder cancer
* spinal cord lesions
* multiple sclerosis
* pelvic radiation
* interstitial cystitis
* artificial sphincter implant
* expected to have changes in medications/doses during the trial
* medically unstable
* Patients with factors that could cause transient UI [e.g., current urinary tract infection (UTI), acute confusion] will be treated in concert with the subject's primary care provider and considered for enrollment if their UI persists.
* conditions that require endocarditis prophylaxis (such as heart valve problems or bacterial endocarditis)

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women over 60 years
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Werner Schaaefer, DI, Principal Investigator — University of Pittsburgh
Locations (1):
- Geriatric Continence Research Unit, NE547 Montefiore UPMC, Pittsburgh, Pennsylvania, United States